CLINICAL TRIAL: NCT00413803
Title: Comparison of Four and Eight Hours Dialysis Sessions in Thrice Weekly Hemodialysis: Long Dialysis Study
Brief Title: Comparison of Four and Eight Hours Dialysis Sessions in Thrice Weekly Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Fresenius Medical Care, Fresenius Medical Care
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-5.1/8
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2009-08-04 (Estimated); Status verified 2009-08

CONDITIONS: End-Stage Renal Disease; Hemodialysis
Keywords: Hemodialysis; Nocturnal dialysis; Cardiovascular disease; Quality of Life; left ventricular hypertrophy
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases; Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): Four-hour dialysis session, blood flow rate 300-400 ml/min
  Interventions: Procedure: 4-hour thrice weekly in center hemodialysis
- 2 (Active Comparator): Eight-hours dialysis session, blood flow rate 200-250 ml/min
  Interventions: Procedure: 8-hour thrice weekly in center hemodialysis

INTERVENTIONS:
Procedure: 4-hour thrice weekly in center hemodialysis — conventional hemodialysis
  Arms: 1
Procedure: 8-hour thrice weekly in center hemodialysis — long dialysis
  Arms: 2

SUMMARY:
The investigators hypothesize that an increase in the duration of dialysis session in thrice weekly center hemodialysis may provide better outcome, less morbidity, higher quality of life, lesser requirement of medications, and lower total cost.

DETAILED DESCRIPTION:
The proposed prospective and controlled clinical trial aims to compare 4-hour and 8-hour dialysis sessions in thrice weekly center HD regarding mortality, hospitalization rate, several clinical and laboratory parameters, and total cost. Four hundred and ten HD patients will be taken into the study. The study will last for 12 months. The patients will be placed in two groups:

1. Four-hour dialysis session, blood flow rate 300-400 ml/min
2. Eight-hours dialysis session, blood flow rate 200-250 ml/min

Sample size is estimated with following hypotheses: twelve months duration of follow-up; twelve months survival of the control group 85%; a bilateral alpha risk equal to 5%; an expectation that 12-months survival to be 95% by 8-hours dialysis; a 85% power to detect the decrease in annual mortality by 8-hours dialysis comparing to 4-hours dialysis; a 10% of dropout rate. The required sample is total 410 patients.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18-years
* On maintenance bicarbonate HD scheduled thrice weekly 12 hours/week; achieved mean single pool Kt/V above 1.2
* Willingness to participate in the study with a written informed consent

Exclusion Criteria:

* To be scheduled for living donor renal transplantation
* To have serious life-limiting co-morbid situations, namely active malignancy, active infection, end-stage cardiac, pulmonary, or hepatic disease
* Pregnancy or lactating
* Current requirement for HD more than three times per week due to medical comorbidity
* GFR greater than 10 ml/min/1.73 m2 as measured by the average of urea and creatinine clearances obtained from a urine collection of at least 24 hours
* Use of temporary catheter
* Current use of investigational drugs or participation in an interventional clinical trial that contradicts or interferes with the therapies or measured outcomes in this trial
* Mental incompetence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
total mortality | one year

SECONDARY OUTCOMES:
cardiovascular mortality | one year
changes in health-related quality of life, depression burden, cognitive function | one year
required medications | one year
total cost | one year
changes in blood pressure, left ventricular geometry, coronary artery calcification, arterial stiffness,upper mid-arm circumference,hematocrit and related rHu-EPO doses, the levels of phosphorus, albumin, lipid parameters, hsCRP, and β-2 microglobulin | one year
hospitalization rate | one year
Vascular access patency | one year
post-dialysis body weight and total body water | one year
arrythmia episodes determined by Holter-ECG | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ercan Ok, MD, Principal Investigator — Ege University
Locations (2):
- Turkey (Türkiye) (2):
  - FMC Turkey Clinics, Adana
  - Ege University School of Medicine Nephrology Department, Izmir

REFERENCES:
- [Derived] Demirci MS, Celik G, Ozkahya M, Tumuklu M, Toz H, Asci G, Duman S, Basci A, Kircelli F, Ozdogan O, Demirci C, Can L, Isik IO, Ok E; Long Dialysis Group. Effects of thrice weekly nocturnal hemodialysis on arterial stiffness. Atherosclerosis. 2012 Feb;220(2):477-85. doi: 10.1016/j.atherosclerosis.2011.11.015. Epub 2011 Nov 19. PMID 22172590